CLINICAL TRIAL: NCT03546868
Title: Phase 2, Open-label, Non-randomized, Single Center Study to Explore Diagnostic Validity of [18F]FSPG PET for the Assessment of Disease Activity in Subjects With Inflammatory Bowel Disease.
Brief Title: Diagnostic Validity of [18F]FSPG PET for the Assessment of Disease Activity in Inflammatory Bowel Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FSPG -1701
Record Dates: First submitted 2018-05-10; First posted 2018-06-06 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease | interventions — 4-(3-fluoropropyl)glutamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ulcerative Colitis (Experimental): Patients with ulcerative colitis undergoing [18F]FSPG PET/CT scan
  Interventions: Drug: [18F]FSPG
- Crohn's disease (Experimental): Patients with Crohn's disease undergoing [18F]FSPG PET/CT scan
  Interventions: Drug: [18F]FSPG

INTERVENTIONS:
Drug: [18F]FSPG — Patients will receive 200 MBq of [18F]FSPG and undergo PET/CT for assessing disease activity in inflammatory bowel disease
  Other Names: FSPG

SUMMARY:
Diagnostic validity of [18F]FSPG for assessing disease activity will be assessed in subjects with inflammatory bowel disease.

DETAILED DESCRIPTION:
[18F]FSPG PET/CT imaging will noninvasively assess system xc- of cancer and inflammation. Diagnostic validity of [18F]FSPG for assessing disease activity will be assessed in subjects with inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject is aged between 19 and 79 years and male or female of any race/ethnicity.
* Subject has had ulcerative colitis or Crohn's disease diagnosed by clinical, endoscopic and histologic evidence at least 3 months prior to screening.
* Subject has symptoms suggestive of active disease at the time of enrollment.
* Subject is scheduled to undergo sigmoidoscopy or colonoscopy for ulcerative colitis or Crohn's disease within 7 days prior to or after the planned study with [18F]FSPG administration.

Exclusion Criteria:

* Subject or subject's legally acceptable representative does not provide written informed consent.
* Subject displays clinical signs of ischemic colitis or has an evidence of pathogenic bowel infection.
* Subject is diagnosed as having inflammatory bowel disease unclassified.
* Subject has been treated with sulfasalazine or intravenous corticosteroids within the previous four weeks prior to the planned study with [18F]FSPG administration.
* Dose escalation of the current inflammatory bowel disease drugs or starting a new oral aminosalicylate, corticosteroid, immunomodulator, biologics, antibiotics, probiotics, or topical preparations is scheduled from the study enrollment to the scheduled sigmoidoscopy or colonoscopy, or 24 hours after [18F]FSPG administration . The dose escalation or starting a new antidiarrheal and/or analgesic drug is allowed.
* Female subject is pregnant or nursing. Exclusion of the possibility of pregnancy is made by one of the following: 1) Woman is physiologically post-menopausal (cessation of menses for more than 2 years), 2) woman is surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy, or 3) if the woman is of childbearing potential, a serum or urine pregnancy test performed within 24 hours immediately prior to administration of [18F]FSPG has to be negative and the women is advised to apply contraceptive measures during her participation in this study.
* Subject has concurrent severe and/or uncontrolled and/or unstable medical disease (e.g. congestive heart failure, acute myocardial infarction, severe pulmonary disease, chronic renal or hepatic disease which could compromise participation in the study) in the judgment of the investigator.
* Subject is a relative of the investigator, student of the investigator or otherwise dependent.
* Subject has received any investigational drugs or devices within four weeks prior to the study enrollment.
* Subject has been previously included in this study.
* Subject has any other condition or personal circumstances that, in the judgment of the investigator, might make collection of complete data difficult or impossible.
* Subject is allergic to hyoscine or any of ingredients of hyoscine butylbromide, or has myasthenia gravis, megacolon, closed angle glaucoma, or obstructive prostatic hypertrophy.

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-11 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of active disease | 60 - 75 min
  Sensitivity and specificity of [18F]FSPG PET/CT for the diagnosis of subjects with endoscopic evidence of active disease
Sensitivity and specificity of severe disease (presence of ulceration) | 60 - 75 min
  Sensitivity and specificity of [18F]FSPG PET/CT for the diagnosis of subjects with endoscopic evidence of severe disease (presence of ulceration)

SECONDARY OUTCOMES:
Area under the receiver operating characteristic curve of active disease | 60 - 75 min
  Area under the receiver operating characteristic curve, sensitivity and specificity of segmental [18F]FSPG PET/CT assessment for detecting bowel segments with endoscopic evidence of active disease

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Asan Foundation, Seoul, Songpa-gu
  - Asan Foundation, Seoul

IPD SHARING:
Plan to Share IPD: Undecided